CLINICAL TRIAL: NCT03694067
Title: Assessment of the Role of the JAK-STAT Pathway in the Pathogenesis of Male Androgenetic Alopecia
Brief Title: Androgenetic Alopecia and the JAK-STAT Pathway
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya AlOrbani, Lecturer of Dermatology, Cairo University
Other Study IDs: Atm567
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Androgenetic Alopecia
Keywords: Androgenetic; Alopecia; JAK; STAT
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 1mm punch skin biopsies will be taken to be analyzed by PCR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Androgenetic alopecia patients: Two 1 mm scalp punch skin biopsy will be taken per patient
  Interventions: Other: Punch skin biopsy

INTERVENTIONS:
Other: Punch skin biopsy — One 1 mm punch biopsy will be taken from the patients from balding scalp. Another 1 mm punch biopsy will be taken from an area of occipital non-balding scalp of the same individual. Local anesthesia will be injected around the biopsy site beforehand.

SUMMARY:
It is a well known fact that the JAK-STAT pathway plays a pivotal role in the pathogenesis of alopecia areata. Both phosphorylated STAT 1 and 3 have been found to be upregulated in the disease. However, whether this pathway plays a role in other hair loss disorders remains unclear. The study aims at assessing STAT3 levels in male patients with androgenetic alopecia. The investigators hypothesize that STAT3 levels will be elevated (due to a previous study proving that JAK-STAT pathway is involved in non-immune mediated hair loss in mice.

DETAILED DESCRIPTION:
Background and rationale Androgenetic alopecia occurs in men and women,and is characterised by the loss of hair from the scalp in a defined pattern. Determining factors appear to be genetic predisposition coupled with the presence of sufficient circulating androgen.

The transformation of testosterone into dihydrotestosterone(DHT) by type 2 5-alpha reductase, which causes hair miniaturization,is universally accepted as the main player in the disease's pathogenesis. Nonetheless,how DHT causes hair thinning is not well understood. New studies revealed that a lymphocytic microfolliculitis targeting the bulge epithelium along with deposits of epithelial basement membrane zone immunoreactants are frequent findings in androgenetic alopecia and could point toward an immunologically driven trigger.

Tyrosine kinases (TKs) are enzymes involved in intracellular signaling that catalyze the phosphorylation of tyrosine residues on protein substrates. They are key components of signaling pathways that drive any array of cellular responses including proliferation, differentiation, migration and survival. Janus kinases (JAKs) are specific TKs.

Signal transducer and activator of transcription (STAT) proteins are transcription factorsprimarily phosphorylated and activated by JAKs.The JAK-STAT pathway is utilized by cytokines including interleukins (ILs), interferons (IFNs), and other molecules to transmit signals from the cell membrane to the nucleus. Growing evidence suggests that JAK inhibitors are efficacious in atopic dermatitis, alopecia areata, psoriasis and vitiligo.

It is a well known fact that the JAK-STAT pathway plays a pivotal role in the pathogenesis of alopecia areata. Both phosphorylated STAT 1 and 3 have been found to be upregulated in the disease. However, whether this pathway plays a role in other hair loss disorders remains unclear. A study showedthat topical treatment of mouse and human skin with small molecule inhibitors of the JAK-STATpathway resulted in rapid onset of anagen and subsequent hair growth. It was shown that JAK inhibition regulates the activation of key hair follicle populations such as the hair germ. These findings indicate that the JAK-STAT pathway may be involved, not only in immune-mediated hair loss (alopecia areata), but also in the normal hair cycle.

This current study aims at assessing STAT3 levels in patients with androgenetic alopecia, in an attempt to detect a possible role of the JAK-STAT pathway in the pathogenesis of the disease.

Objective:

The objective is to compare tissue levels of STAT3 in androgen-dependant areas in male androgenetic alopecia patients with their level in non-involved, non-androgen dependant areas (occipital scalp) in the same subjects.

Population of study & disease condition (e.g women with hepatitis, ............) Males with androgenetic alopecia

Background and demographic characteristics( e.g age,.......)

* Age above 18 years.
* Males

Interventions :

Each subject will be subjected to:

* Informed consent.
* Detailed history and clinical evaluation to determine severity of disease.
* Punch biopsies (1mm) of affected area of scalp (androgen dependent area) from 25 patients with androgenetic alopecia.
* Punch biopsies(1mm) of normal area of scalp from occipital scalp (non-androgen dependent area) from the same 25 patients
* Quantification of STAT3 by polymerase chain reaction (PCR).

Sample size (number of participants included)

* 25 participants (That will serve as both patients and controls)
* Sample size calculation was done using G ⃰ Power 3.1.9.2.

Possible. Risk Bleeding, secondary infection, scarring.

ELIGIBILITY:
Inclusion Criteria:

* Males with androgenetic alopecia not receiving topical treatment nor systemic treatment for hair loss for at least 6 month prior to the study

Exclusion Criteria:

* Patients with localized or generalized hair loss due to causes other than androgenetic alopecia.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Specialized dermatology clinic at Cairo University
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Different in STAT3 | 6 months
  STAT3 levels in androgen-dependant areas compared to non-involved areas from occipital scalp(in an attempt to assess the possible role of the JAK-STAT pathway in androgenetic alopecia).

SECONDARY OUTCOMES:
Correlating STAT3 with severity | 6 months
  The relation of STAT3 levels to the severity of androgenetic alopecia (Hamilton-Norwood scale)

CONTACTS AND LOCATIONS:
Overall Officials: Akmal S Hassan, MD, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Damsky W, King BA. JAK inhibitors in dermatology: The promise of a new drug class. J Am Acad Dermatol. 2017 Apr;76(4):736-744. doi: 10.1016/j.jaad.2016.12.005. Epub 2017 Jan 28. PMID 28139263
- [Background] Ellis JA, Sinclair R, Harrap SB. Androgenetic alopecia: pathogenesis and potential for therapy. Expert Rev Mol Med. 2002 Nov 19;4(22):1-11. doi: 10.1017/S1462399402005112. PMID 14585162
- [Background] Harel S, Higgins CA, Cerise JE, Dai Z, Chen JC, Clynes R, Christiano AM. Pharmacologic inhibition of JAK-STAT signaling promotes hair growth. Sci Adv. 2015 Oct 23;1(9):e1500973. doi: 10.1126/sciadv.1500973. eCollection 2015 Oct. PMID 26601320
- [Background] Magro CM, Rossi A, Poe J, Manhas-Bhutani S, Sadick N. The role of inflammation and immunity in the pathogenesis of androgenetic alopecia. J Drugs Dermatol. 2011 Dec;10(12):1404-11. PMID 22134564
- [Background] O'Shea JJ, Schwartz DM, Villarino AV, Gadina M, McInnes IB, Laurence A. The JAK-STAT pathway: impact on human disease and therapeutic intervention. Annu Rev Med. 2015;66:311-28. doi: 10.1146/annurev-med-051113-024537. PMID 25587654
- [Background] Paniagua RT, Fiorentino DF, Chung L, Robinson WH. Tyrosine kinases in inflammatory dermatologic disease. J Am Acad Dermatol. 2011 Aug;65(2):389-403. doi: 10.1016/j.jaad.2010.04.026. Epub 2010 Jun 26. PMID 20584561
- [Background] Schwartz DM, Bonelli M, Gadina M, O'Shea JJ. Type I/II cytokines, JAKs, and new strategies for treating autoimmune diseases. Nat Rev Rheumatol. 2016 Jan;12(1):25-36. doi: 10.1038/nrrheum.2015.167. Epub 2015 Dec 3. PMID 26633291
- [Background] Rawlings JS, Rosler KM, Harrison DA. The JAK/STAT signaling pathway. J Cell Sci. 2004 Mar 15;117(Pt 8):1281-3. doi: 10.1242/jcs.00963. No abstract available. PMID 15020666
- [Background] Whiting DA. Possible mechanisms of miniaturization during androgenetic alopecia or pattern hair loss. J Am Acad Dermatol. 2001 Sep;45(3 Suppl):S81-6. doi: 10.1067/mjd.2001.117428. PMID 11511857
- [Background] Xing L, Dai Z, Jabbari A, Cerise JE, Higgins CA, Gong W, de Jong A, Harel S, DeStefano GM, Rothman L, Singh P, Petukhova L, Mackay-Wiggan J, Christiano AM, Clynes R. Alopecia areata is driven by cytotoxic T lymphocytes and is reversed by JAK inhibition. Nat Med. 2014 Sep;20(9):1043-9. doi: 10.1038/nm.3645. Epub 2014 Aug 17. PMID 25129481